CLINICAL TRIAL: NCT02512861
Title: Parasternal Nerve Block Using Bupivacaine for Postoperative Analgesia in Children Undergoing Cardiac Surgery: A Prospective: Double-Blind, Randomized Controlled Trial
Brief Title: Parasternal Nerve Block Using Bupivacaine for Postoperative Analgesia in Children Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1311-105
Record Dates: First submitted 2014-06-06; First posted 2015-07-31 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Bupivacaine; Cardiac Surgery; Pediatrics; Nerve Block
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Active Comparator): Bupivacaine as a parasternal nerve block following pediatric cardiothoracic surgery
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine will be administered bilaterally to the parasternal intercostal spaces during surgery according to these doses:
  Under 20kgs weight: 0.25% Bupivacaine at 1 milliliter/kilogram (1ml/kg); Above 20kgs weight: 0.5% Bupivacaine at 0.5 ml/kg up to a maximum of 25ml of 0.5% Bupivacaine for patients > 50 kgs
  Other Names: Marcaine; Sensorcaine
  Arms: Bupivacaine
Drug: Placebo — Saline will be administered bilaterally to the parasternal intercostal spaces during surgery according to these doses:
  Under 20kgs weight: 1 milliliter/kilogram (1ml/kg); Above 20kgs weight: 0.5 ml/kg up to a maximum of 25ml for patients > 50 kgs
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
All pediatric patients who undergo cardiac surgery require analgesic medications for postoperative pain control and many require sedation to facilitate comfort with cares. Parasternal infiltration of local anesthetic for nerve blocks is a simple option to postoperative analgesia. The investigators hypothesize that Bupivacaine, a parasternal nerve block administered in pediatric patients undergoing cardiac surgery will reduce the requirement of Opioids and other pain medications as well as decrease postoperative pain scores. This is a prospective, double-blind, randomized controlled trial. Subjects are randomized to receive either 0.25% Bupivacaine or normal saline following their cardiothoracic surgery.

DETAILED DESCRIPTION:
One of the most challenging struggles in clinical practices in pediatric cardiac intensive care units is the provision of optimal and safe postoperative analgesia and sedation. All pediatric patients who undergo cardiac surgery require analgesic medications for postoperative pain control and many require sedation to facilitate comfort with cares. Parasternal infiltration of local anesthetic for nerve blocks is a simple option to postoperative analgesia. Bupivacaine is a local anesthetic that can be injected into the intercostal spaces on each side of a sternotomy to induce nerve block.

The purpose of this study is to evaluate whether the use of Bupivacaine as a nerve block in children undergoing cardiothoracic surgery will reduce postoperative pain medication use and decrease postoperative pain scores. The investigators hypothesize that the administration of Bupivacaine bilaterally into the posterior intercostal spaces on each side of a sternotomy following cardiothoracic surgery will reduce the requirement of pain medications as well as decrease postoperative pain scores.

This is a prospective, randomized, double-blind, control study. Subjects are randomized into two arms: those who receive 0.25% Bupivacaine and those who receive placebo (normal saline). Subjects receive 1 milliliter per kilogram up to 20 kilograms, then 0.5 milliliters per kilogram up to 50 kilograms of study drug.

Subjects are followed for 5 days postoperatively, then on day of discharge. Pain medication administered and Face, Legs, Activity, Cry, and Consolability (FLACC) scores are recorded daily for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17 years old at time of surgery
* Society of Thoracic Surgeons- European Association for Cardio-Thoracic Surgery (STAT) mortality categories 1-3
* Surgical intervention requiring median sternotomy
* Expected extubation within 24 hours of surgery

Exclusion Criteria:

* Known allergic reaction or hypersensitivity to Bupivacaine or to any local anesthetic agent of the amide type
* Delayed sternum closure

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis X Moga, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine: Bupivacaine as a parasternal nerve block following pediatric cardiothoracic surgery
  Bupivacaine: Bupivacaine will be administered bilaterally to the parasternal intercostal spaces during surgery according to these doses:
  Under 20kgs weight: 0.25% Bupivacaine at 1 milliliter/kilogram (1ml/kg); Above 20kgs weight: 0.5% Bupivacaine at 0.5 ml/kg up to a maximum of 25ml of 0.5% Bupivacaine for patients > 50 kgs
- Placebo: Normal Saline
  Placebo: Saline will be administered bilaterally to the parasternal intercostal spaces during surgery according to these doses:
  Under 20kgs weight: 1 milliliter/kilogram (1ml/kg); Above 20kgs weight: 0.5 ml/kg up to a maximum of 25ml for patients > 50 kgs
Period: Overall Study
Arm/Group | Bupivacaine | Placebo
Started | 44 | 49
Completed | 38 | 40
Not Completed | 6 | 9
Not completed — Protocol Violation | 3 | 7
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Placebo | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1 [0.4 to 3.3] | 0.8 [0.4 to 3.7] | 0.84 [0 to 3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 23 | 22 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 3 | 2 | 5
  White/Caucasian | 30 | 26 | 56
  Asian | 0 | 1 | 1
  Hispanic/Latino | 2 | 2 | 4
  American Indian/Alaskan | 0 | 4 | 4
  Bi-racial | 0 | 1 | 1
  Declined | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 78
Comorbidities [Count of Participants; unit: Participants] — Any additional medical conditions that the patient had in addition to the cardiac defect were collected and categorized into the following:
  1. Respiratory
  2. Gastrointestinal
  3. Genetic
  4. Neurodevelopmental/Developmental Delay
  5. Other
  Participants
    Respiratory | 0 | 3 | 3
    Gastrointestinal | 1 | 1 | 2
    Genetic | 11 | 7 | 18
    Neurodevelopmental/Developmental Delay | 1 | 2 | 3
    None | 24 | 25 | 49
    Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Fentanyl/Equivalent Day 0-1
Time Frame: Day of Surgery and Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: mcg/kg/day
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 38 | 40
mcg/kg/day | 23.6 [10.7 to 34.3] | 22.4 [13.3 to 32.6]

2. Primary Outcome: Patient-Controlled Analgesia (PCA) Fentanyl/Equivalent Day 0-1
Time Frame: Day of Surgery and Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: mcg/kg/day
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 38 | 40
mcg/kg/day | 15.7 [8.5 to 22.1] | 14.6 [10.6 to 21.7]

3. Secondary Outcome: Postoperative Length of Intubation
Time Frame: 5 days post cardiac surgery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 38 | 40
hours | 5.9 [3.7 to 19.5] | 6.4 [3.3 to 22.1]

4. Secondary Outcome: Postoperative Cortisol Levels
Time Frame: 12 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: microgram/deciliter
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 38 | 40
microgram/deciliter | 25.4 [15.5 to 44.8] | 27.7 [14.9 to 59.4]

5. Secondary Outcome: Postoperative Pain Scores-Face, Legs, Activity, Cry, Consolability (FLACC) Scale
Description: Face, Legs, Activity, Cry, Consolability (FLACC) scale: range is from 0 to 10 and a higher score indicates greater level of pain (worse outcome).
Time Frame: Day of Surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 24 | 28
score on a scale | 0 [0 to 2.88] | 0 [0 to 1.15]

6. Secondary Outcome: Postoperative Pain Scores-State Behavioral Scale (SBS)
Description: State Behavioral Scale (SBS): range is from -3 to 2. A higher score indicates a patient is more uncomfortable and agitated (worse outcome).
Time Frame: Day of Surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 24 | 28
score on a scale | -0.25 [-1 to 1] | -0.25 [-1 to 0]

7. Secondary Outcome: Postoperative Cortisol Levels
Time Frame: 36 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: microgram/deciliter
Arm/Group | Bupivacaine | Placebo
Number analyzed (Participants) | 38 | 40
microgram/deciliter | 9.4 [5.1 to 17.3] | 9.1 [3.6 to 20.7]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the first five post-operative days.
Description: The method for collecting adverse event information was via daily collection form/questionnaire by the study coordinator for the first five post-operative days.
Arm/Group | Bupivacaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 3/38 | 6/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine (N=38) | Placebo (N=40)
Shallow Breathing/Increased Work of Breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Patient required either non-invasive respiratory support or reintubation
Significant blood/chest tube losses requiring transfusion or fluid resuscitation (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Pneumothorax or Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Patient required reinitiation of chest tubes
Acute respiratory syncytial virus leading to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes